CLINICAL TRIAL: NCT02417168
Title: Procalcitonin Levels as a Predictor of Bacteremia in Febrile Pediatric Oncology Patients - Pilot Study
Brief Title: Procalcitonin Levels as a Predictor of Bacteremia in Febrile Pediatric Oncology Patients-Pilot Study
Status: Terminated | Type: Observational
Why Stopped: PI left study site
Sponsor: CAMC Health System (Other)
Collaborators: CureSearch for Children's Cancer (Unknown)
Responsible Party: Sponsor
Other Study IDs: 14-42
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Cancer; Bacteremia
MeSH Terms: conditions — Neoplasms; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fevers raise the concern for serious bacterial infections in pediatric oncology patients receiving chemotherapy. The gold standard for diagnosing bacteremia (bacterial infection of the blood) is a blood culture. However, bacterial growth may not occur for 48 hours or there can be a false negative result.

Thus, the biomarker, procalcitonin, has been investigated for its predictive ability to identify bacteremia earlier than blood culture. We believe that procalcitonin can assist in differentiating bacteremia from non-bacteremia infections in febrile pediatric oncology patients. A reliable predictor of bacteremia infections in pediatric oncology patients should decrease hospitalizations for fever and unnecessary antibiotic treatment.

In our study we will measure procalcitonin levels in pediatric oncology patients presenting with fever. We will measure procalcitonin at the time of admission which is part of our standard of care for febrile pediatric oncology admissions. For the purpose of our study, we will additionally measure procalcitonin levels at 12 hours and at 24 hours post admission. We will examine procalcitonin levels at these three timepoints to determine if elevated procalcitonin levels predict bacteremia in pediatric oncology patients with and without neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of birth to seventeen years.
* Present to Charleston Area Medical Center Women and Children's Hospital
* Existing pediatric oncology diagnosis.
* Temperature greater than 38.0 C or 100.5 Fahrenheit.
* Central venous access or functional port available.

Exclusion Criteria:

* Any non-pediatric (eighteen years and above) oncology patient or a non-oncology patient.
* The patient does not have central venous access or a port from which the blood can be drawn.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between the ages of birth to seventeen years who have an existing oncologic diagnosis and who present with fever to Charleston Area Medical Center Women and Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Change in procalcitonin levels | 24 hours
  Procalcitonin will be measured at the time of admission (Zero hours) and at 12, at 24 hours from admission.

SECONDARY OUTCOMES:
The presence of bacteremia | 1 week
  Blood will be cultured for bacteria

CONTACTS AND LOCATIONS:
Locations (1):
- CAMC Health Systems, Charleston, West Virginia, United States